CLINICAL TRIAL: NCT07157813
Title: Improving Lifestyle Habits and Metabolic Health in Forensic Psychiatric Patients
Acronym: FOR-HEALTH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOR-HEALTH; 2025-02066-01 (Other: The Swedish Ethical Review Authority)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Forensic Psychiatric Patients; Cardio Vascular Disease; Health Promotion; Forensic Mental Health; Forensic Psychiatry; Physical Fittness; Diet Habits; Smoking Cessation
Keywords: Health dialog
MeSH Terms: conditions — Feeding Behavior; Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Health Dialogue (Experimental): Participants receive two nurse-led Structured Health Dialogue sessions in addition to usual care. Each session includes a standardized health screening, blood sampling, and physiological measurements, together with a structured discussion tailored to the individual's risk profile. The dialogues and questionnaires are conducted at baseline and at 12 months. At 6 months, only blood sampling, questionnaires and measurements are repeated (no dialogues).
  Interventions: Behavioral: Structured Health Dialogue
- Control group (No Intervention): Participants receive usual care. They undergo blood sampling, physiological measurements, and questionnaires at baseline, 6 months and at 12 months. Participants in the control group do not receive any Structured Health Dialogue sessions.

INTERVENTIONS:
Behavioral: Structured Health Dialogue — In addition to usual care, participants take part in two nurse-led Structured Health Dialogue (SHD) sessions at baseline and 12 months. The results from the measurements and questionnaires are integrated into an individualized visual risk profile ("health curve"). This profile is used as the foundation for a 60-90 minute dialogue, guided by motivational interviewing principles, to enhance risk awareness, promote self-reflection, and support participants in setting achievable goals for lifestyle improvement.
  Arms: Structured Health Dialogue

SUMMARY:
Background:People in compulsory forensic psychiatric care experience high rates of metabolic syndrome, cardiovascular disease, and related lifestyle risk factors, yet structured preventive health interventions are uncommon in secure psychiatric settings. The Structured Health Dialogue (SHD), a Swedish primary care model for cardiovascular disease prevention, combines motivational interviewing with individualised risk assessment and tailored lifestyle advice.

Objective:To evaluate the feasibility, acceptability, and preliminary effects of an adapted SHD intervention in forensic psychiatric inpatient care.

Methods:This single-centre, parallel-group, randomized controlled feasibility trial will recruit 50 adults aged 18-64 years from a secure forensic psychiatric clinic in Sweden. Participants will be randomized (1:1) to SHD plus usual care or usual care alone. The SHD includes health screening, lifestyle assessment, personalised cardiovascular risk feedback, and tailored recommendations. Primary outcomes are recruitment, retention, dropout, and assessment completion rates. Secondary outcomes include changes in metabolic risk factors and patient-reported quality of life and functioning (EQ-5D-5L, Mental Fatigue Scale) from baseline to 12 months.

Conclusion: This study will inform the feasibility and potential effectiveness of implementing structured, person-centred preventive health interventions in forensic psychiatric care, guiding the design of a future full-scale trial.

DETAILED DESCRIPTION:
Individuals receiving compulsory forensic psychiatric care typically present with severe mental disorders such as schizophrenia, schizoaffective disorder, or personality disorders, and are legally detained following offenses committed under the influence of psychiatric illness. This patient population has a markedly reduced life expectancy-by up to 15-20 years-primarily due to preventable somatic conditions such as cardiovascular disease, type 2 diabetes, and other metabolic disorders. Contributing factors include sedentary lifestyle, unhealthy dietary patterns, tobacco and alcohol use, limited health literacy, and the metabolic side effects of long-term antipsychotic treatment. The restrictive environment of secure psychiatric care may further limit opportunities for physical activity and healthy eating. Epidemiological studies consistently show that obesity, metabolic syndrome, and cardiometabolic risk factors are highly prevalent among forensic psychiatric inpatients, with rates often exceeding those observed in both the general population and other psychiatric settings. Despite this, structured preventive health interventions are rarely implemented in forensic psychiatry, and evidence on how such programs can be adapted to this context remains limited.

The Structured Health Dialogue (SHD) is a validated Swedish primary care method for cardiovascular disease prevention. It integrates evidence-based behavioural strategies such as motivational interviewing with an individualized risk assessment. Central to the method is a visual tool, the so-called "health curve," which is generated from systematically collected data including biometric measurements, laboratory tests, and a structured lifestyle questionnaire. This visual risk profile provides a concrete and accessible summary of the individual's cardiometabolic risk factors, which is then used as the foundation for the health dialogue. By combining objective data with motivational interviewing, SHD facilitates patient engagement, enhances understanding of risk, and supports goal-setting for behavioural change. Evidence from primary care indicates that SHD improves lifestyle habits, metabolic health indicators, and patient participation in preventive care. However, its feasibility and potential effectiveness in compulsory forensic psychiatric care have not yet been evaluated in a randomized controlled setting.

This study is designed as a single-centre, parallel-group randomized controlled feasibility trial conducted at the Regional Forensic Psychiatric Clinic in Växjö, Sweden. The trial follows methodological guidance for feasibility and pilot studies and will be reported according to the CONSORT 2010 extension for pilot and feasibility trials. Eligible participants will be randomized in a 1:1 ratio to either the intervention group (SHD plus usual care) or the control group (usual care only). Randomization will be stratified by ward type and implemented using a computer-generated sequence with block randomization within security classes I-III. Block randomization is applied to ensure balance between groups, as patients in class I wards are often in an earlier phase of treatment or present with more severe psychiatric symptoms compared to patients in classes II and III. From a methodological perspective, stratification and block randomization by security class reduces the risk of systematic imbalance in baseline characteristics, thereby controlling for potential confounding related to ward type and severity of illness.

The intervention consists of two nurse-led SHD sessions delivered over a 12-month period. Each session lasts approximately 60-90 minutes and includes systematic health screening (anthropometric and biometric measures, fasting blood tests), a structured lifestyle questionnaire, and individualized risk feedback using the health curve. The sessions employ motivational interviewing techniques to support patient autonomy, set realistic lifestyle goals, and identify strategies for behavioural change. Tailored recommendations and referrals to relevant health services are provided when needed.

Assessments are scheduled at baseline, 6 months, and 12 months, including biometric measurements and validated self-report questionnaires on lifestyle behaviours, quality of life, and functioning. Feasibility outcomes include recruitment rates, retention, adherence to intervention and follow-up, and completeness of data collection. Secondary outcomes will provide preliminary estimates of intervention effects on metabolic risk factors, lifestyle habits, and self-reported quality of life, which will inform the design of a future adequately powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64 years
* Hospitalized at the forensic psychiatric clinic in Växjö, Sweden.

Exclusion Criteria:

* Severe language barriers.
* Severe cognitive impairment
* Acute psychiatric states (e.g., suicidality or acute psychosis)
* Aggression hindering safe participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study design and Targeted health dialogue | 24-month
  Recruitment rate in both groups calculated continuously throughout the recruitment period, reported as the number of participants enrolled per month.
Feasibility of the study design and Targeted health dialogue | 24-month
  Dropout rate in both groups calculated continuously throughout the study period, reported as the proportion of participants who discontinue participation before completion of follow-up.

SECONDARY OUTCOMES:
Biometric measures, Body Mass Index (BMI) | 12 months
  Calculated in both groups at baseline, 6 months, and 12 months from measured body weight and height using standard clinical equipment and protocols. Category BMI Range (kg/m²) Underweight < 18.5 Normal weight 18.5 - 24.9 Overweight 25.0 - 29.9 Obesity Class I 30.0 - 34.9 Obesity Class II 35.0 - 39.9 Obesity Class III (severe) ≥ 40.0 In the "Hälsokurvan" system, the cut-off values for BMI differ from the standard WHO categories. For men, a BMI below 27.0 is classified as low risk (green), 27.0-36.9 as moderate risk (yellow), and 37.0 or higher as high risk (orange). For women, a BMI below 29.0 is considered low risk, 29.0-38.9 moderate risk, and 39.0 or higher high risk.
Biometric measures, Waist-to-Hip Ratio | 12 months
  Measured in both groups at baseline, 6 months, and 12 months using a measuring tape according to standard procedures. n the "Hälsokurvan" system, waist-to-hip ratio (WHR) is divided into four risk categories. For men, values below 0.90 are classified as low risk, 0.90-0.94 as moderate risk, 0.95-0.99 as high risk, and 1.00 or higher as very high risk. For women, values below 0.78 are classified as low risk, 0.78-0.82 as moderate risk, 0.83-0.87 as high risk, and 0.88 or higher as very high risk.
Biometric measures, Blood Pressure | 12 months
  Recorded in both groups at baseline, 6 months, and 12 months using standard clinical procedures. In the "Hälsokurvan" system, normal blood pressure is defined as systolic ≤130 mmHg and/or diastolic ≤85 mmHg in otherwise healthy individuals. Values above this level are categorized into increasing risk levels: systolic 140-169 mmHg or diastolic 90-104 mmHg corresponds to a moderate (yellow) category, 170-199/105-114 mmHg to a high (orange) category, and systolic ≥200 mmHg or diastolic ≥115 mmHg to a very high (red) category.
Biometric measures, Fasting Plasma Glucose | 12 months
  Measured in both groups at baseline, 6 months, and 12 months through blood sampling under standardized conditions. Both short-term fP-Glucose (mmol/L) and long-term glucose HbA1c (mmol/mol) control will be assessed.
Biometric measures, Blood Lipid Status | 12 months
  Assessed in both groups at baseline, 6 months, and 12 months via blood sampling under standardized conditions, including total cholesterol (mmol/L), LDL(mmol/l), HDL(mmol/L), and triglycerides (mmol/L). In the Hälsokurvan system, blood lipids are primarily assessed through total cholesterol. Total cholesterol values below 7.5 mmol/L and LDL values below 4.9 mmol/L are managed by calculating the SCORE risk to classify overall cardiovascular risk.
  The system classifies risk into four levels (green, yellow, orange, red) based on these thresholds together with additional risk factors.
Biometric measurments, Body Weight | 12 months
  Measured (kg) in both groups at baseline, 6 months, and 12 months using a calibrated clinical scale according to standard procedures.
Biometric measures, Body Length (Height) | 12 months
  Measured (cm) in both groups at baseline using a stadiometer according to standard clinical equipment and protocols.
Lifestyle Habits - Physical Activity | 12 months
  Categorised according to the Hälsokurvan health survey standard. Measured in both groups at baseline and 12 months.
  Green (low risk): ≥2000 kcal/week or ≥300 min/week (≥10,000 steps/day) Yellow (moderate risk): 1000-1999 kcal/week or 150-299 min/week Orange (high risk): 500-999 kcal/week or 60-149 min/week Red (very high risk): <500 kcal/week or <60 min/week Outcome: Improvement = one-step reduction in risk from baseline.
Lifestyle Habits - Diet | 12 months
  Categorised according to the Hälsokurvan health survey standard.Measured in both groups at baseline and 12 months.
  Green (low risk): Healthy diet in line with national recommendations (high in fruit/vegetables, whole grains, legumes, fish; low in salt, sugar, red/processed meat) Yellow (moderate risk): Partly healthy diet with clear areas for improvement Orange (high risk): Several unhealthy components (high sugar, saturated fat, processed meat) Red (very high risk): Predominantly unhealthy diet (energy-dense, nutrient-poor, minimal fruit/vegetables) Outcome: Improvement = one-step reduction in risk from baseline
Lifestyle Habits - Tobacco Use | 12 months
  Categorised according to the Hälsokurvan health survey standard.Measured in both groups at baseline and 12 months.
  Green (low risk): No tobacco or nicotine use Yellow (moderate risk): Former or occasional user (non-daily) Orange (high risk): Daily use in small amounts (e.g., 1-9 cigarettes/day) Red (very high risk): Daily use in larger amounts (≥10 cigarettes/day or equivalent) Outcome: Improvement = one-step reduction in risk from baseline
Lifestyle Habits - Alcohol Consumption | 12 months
  Categorised according to the Hälsokurvan health survey standard.Measured in both groups at baseline and 12 months.
  Green (low risk): <4 standard drinks/week Yellow (moderate risk): 4-9 drinks/week Orange (high risk): 10-18 drinks/week or binge ≥4 drinks/monthly Red (very high risk): >18 drinks/week or binge ≥4 drinks/weekly Outcome: Improvement = one-step reduction in risk from baseline
Mental Fatigue | 12 months
  Change in Mental Fatigue Scale (MFS) total score from baseline to 12 months. The MFS ranges from 0 (no mental fatigue) to 42 (maximum mental fatigue). Higher scores indicate worse outcome (greater fatigue), while lower scores indicate better outcome (less fatigue).
Self-Reported Health Status | 12 months
  Change in health status from baseline to 12 months measured with the EQ-5D questionnaire.
  EQ-5D Index score: 0 (equivalent to death) to 1 (full health), higher scores = better outcome.
  EQ-5D VAS: 0 (worst imaginable health) to 100 (best imaginable health), higher scores = better outcome.

OTHER OUTCOMES:
Family History of Cardiovascular Disease and Diabetes | Baseline (single assessment)
  Collected in both groups at baseline through patient interview or from medical records.
Sociodemographic and Clinical Information | Baseline (single assessment)
  Collected in both groups at baseline from patients' medical records, including age, educational level, and current psychiatric diagnoses.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Forensic Psychiatric Clinic, Växjö, Vaxjo, Kronoberg County, Sweden

REFERENCES:
- [Background] Wei TQ, Chu VP, Craig AR, Duffy JE, Obzansky DM, Kilgore D, Masulli IS, Sanders CM, Thompson JC. Automated homogeneous immunoassay for gentamicin on the dimension clinical chemistry system. Clin Chem. 1999 Mar;45(3):388-93. PMID 10053040
- [Background] Cooper A. Hodgkin's disease. Lancet. 1982 Mar 13;1(8272):612-3. No abstract available. PMID 6121193
- [Background] Kuczynska-Sicinska J. [Nephrologic problems in pregnancy]. Pol Arch Med Wewn. 1973 Feb;50(2):221-6. No abstract available. Polish. PMID 4691769
- [Background] Pincelli C, Magni R, Motolese A. Pigmented contact dermatitis from deodorant. Contact Dermatitis. 1993 May;28(5):305-6. doi: 10.1111/j.1600-0536.1993.tb03447.x. No abstract available. PMID 8365140
- [Background] Davis RH, Hynes LV, Eversole-Cire P. Nonsense mutations of the ornithine decarboxylase structural gene of Neurospora crassa. Mol Cell Biol. 1987 Mar;7(3):1122-8. doi: 10.1128/mcb.7.3.1122-1128.1987. PMID 2951589
- [Background] Gupta MM, Srinivasa H, Bhat P. Seroepidemiology of malaria in Karnataka State: longitudinal study of a population from an area with high incidence at Kolar, South India. J Infect Dis. 1983 Sep;148(3):609. doi: 10.1093/infdis/148.3.609. PMID 6352829
- [Background] Hamilton RL, Brown WJ. Medium to aid identification of Serratia marcescens. Am J Med Technol. 1972 Mar;38(3):73-6. No abstract available. PMID 4560167
- [Background] Hsu SH, Pollard MK, Chan MM, Bias WB. Genetic heterogeneity of DR4 in the Old Order Amish and two new HLA-D specificities. Hum Immunol. 1981 Mar;2(2):165-72. doi: 10.1016/0198-8859(81)90063-x. PMID 6167556
- [Background] Winkelmann U. [Influencing factors in the planning of job needs]. Krankenpfl J. 1980 Jul 15;18(7):28-9. No abstract available. German. PMID 6901922
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Johansson B, Starmark A, Berglund P, Rodholm M, Ronnback L. A self-assessment questionnaire for mental fatigue and related symptoms after neurological disorders and injuries. Brain Inj. 2010 Jan;24(1):2-12. doi: 10.3109/02699050903452961. PMID 20001478
- [Background] Uhrskov Sorensen L, Bengtson S, Lund J, Ibsen M, Langstrom N. Mortality among male forensic and non-forensic psychiatric patients: matched cohort study of rates, predictors and causes-of-death. Nord J Psychiatry. 2020 Oct;74(7):489-496. doi: 10.1080/08039488.2020.1743753. Epub 2020 Apr 4. PMID 32248726
- [Background] Dronavalli M, Page A, Ferdousi S, Osaghae M, Sperandei S. Improving metabolic risk in patients with mental illness through 'mental health care plans' in primary health care. Aust N Z J Psychiatry. 2025 Aug;59(8):692-701. doi: 10.1177/00048674251337030. Epub 2025 May 13. PMID 40356373
- [Background] Vorstenbosch EC, Bouman YH, Braun PC, Bulten EB. Psychometric properties of the forensic inpatient quality of life questionnaire: quality of life assessment for long-term forensic psychiatric care. Health Psychol Behav Med. 2014 Jan 1;2(1):335-348. doi: 10.1080/21642850.2014.894890. Epub 2014 Mar 19. PMID 25750786
- [Background] Schel SH, Bouman YH, Vorstenbosch EC, Bulten BH. Development of the forensic inpatient quality of life questionnaire: short version (FQL-SV). Qual Life Res. 2017 May;26(5):1153-1161. doi: 10.1007/s11136-016-1461-9. Epub 2016 Nov 22. PMID 27878427
- [Background] Lingfors H, Persson LG, Lindstrom K, Bengtsson C, Lissner L. Effects of a global health and risk assessment tool for prevention of ischemic heart disease in an individual health dialogue compared with a community health strategy only results from the Live for Life health promotion programme. Prev Med. 2009 Jan;48(1):20-4. doi: 10.1016/j.ypmed.2008.10.009. Epub 2008 Nov 1. PMID 19013188
- [Background] Eliasson M, Eriksson M, Lundqvist R, Wennberg P, Soderberg S. Comparison of trends in cardiovascular risk factors between two regions with and without a community and primary care prevention programme. Eur J Prev Cardiol. 2018 Nov;25(16):1765-1772. doi: 10.1177/2047487318778349. Epub 2018 May 30. PMID 29846119
- [Background] Weinehall L, Hellsten G, Boman K, Hallmans G, Asplund K, Wall S. Can a sustainable community intervention reduce the health gap?--10-year evaluation of a Swedish community intervention program for the prevention of cardiovascular disease. Scand J Public Health Suppl. 2001;56:59-68. PMID 11681565
- [Background] Casey DE, Haupt DW, Newcomer JW, Henderson DC, Sernyak MJ, Davidson M, Lindenmayer JP, Manoukian SV, Banerji MA, Lebovitz HE, Hennekens CH. Antipsychotic-induced weight gain and metabolic abnormalities: implications for increased mortality in patients with schizophrenia. J Clin Psychiatry. 2004;65 Suppl 7:4-18; quiz 19-20. No abstract available. PMID 15151456
- [Background] Laursen TM, Nordentoft M, Mortensen PB. Excess early mortality in schizophrenia. Annu Rev Clin Psychol. 2014;10:425-48. doi: 10.1146/annurev-clinpsy-032813-153657. Epub 2013 Dec 2. PMID 24313570
- [Background] Osby U, Correia N, Brandt L, Ekbom A, Sparen P. Mortality and causes of death in schizophrenia in Stockholm county, Sweden. Schizophr Res. 2000 Sep 29;45(1-2):21-8. doi: 10.1016/s0920-9964(99)00191-7. PMID 10978869
- [Background] Pedersen ALW, Lindekilde CR, Andersen K, Hjorth P, Gildberg FA. Health behaviours of forensic mental health service users, in relation to smoking, alcohol consumption, dietary behaviours and physical activity-A mixed methods systematic review. J Psychiatr Ment Health Nurs. 2021 Jun;28(3):444-461. doi: 10.1111/jpm.12688. Epub 2020 Oct 11. PMID 32916759
- See also: National Strategy for Mental Health and Suicide Prevention — https://www.folkhalsomyndigheten.se/livsvillkor-levnadsvanor/psykisk-halsa-och-suicidprevention/nationell-strategi-for-psykisk-halsa-och-suicidprevention/
- See also: Integrating primary care in a specialized forensic psychiatric setting: predictors of program adherence — https://doi.org/10.1007/s44250-025-00175-0
- See also: Factors associated with quality of life in a cohort of forensic psychiatric in-patients — https://doi-org.ludwig.lub.lu.se/10.1108/14636646200800002